CLINICAL TRIAL: NCT02622477
Title: Clinical Course of Treatment With ESBRIET in Patients With Mild to Moderate IPF
Brief Title: Clinical Progression of Mild to Moderate Idiopathic Pulmonary Fibrosis (IPF) Under a Therapy With Esbriet® (Pirfenidone)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: InterMune Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30016
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Participants with idiopathic pulmonary fibrosis: Participants with idiopathic pulmonary fibrosis receiving Pirfenidone will be observed for treatment responses.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — This is an observational study. Pirfenidone is available as an 267 mg capsule for oral administration.

SUMMARY:
The purpose of the study was to assess the clinical outcome of patients with a mild to moderate IPF after a one-year therapy with Esbriet® (Pirfenidone).

ELIGIBILITY:
Inclusion Criteria:

Adult patients with confident diagnosis of mild to moderate IPF, who had previously not yet been treated with Pirfenidone

Exclusion Criteria:

Hypersensitivity to the active substance or one of the other excipients of Pirfenidone Concomitant use of Fluvoxamin Severe hepatic impairment or end stage liver disease Severe renal impairment (Creatinine-Clearance <30 ml/min) or end stage renal disease requiring dialysis Simultaneous participation in interventional studies Previously treated with Pirfenidone for longer than 30 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with diagnosis of mild to moderate idiopathic pulmonary fibrosis (IPF), who had previously not yet been treated with Pirfenidone
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Categorical Decrease Of The Vital Capacity And Forced Volume Capacity (>= 5 % Respectively 10% Compared To The Previous Examination Findings) Under Treatment | -3 to 8 months before inclusion, appointment 0, and 3, 6, 9 and 12 months after appointment
Categorical Decrease of the 6-Minute Walking Distance (>= 50 Metres Compared to the Previous Examination Findings) Under Treatment | Appointment 0, and 3, 6, 9 and 12 months after appointment 0
Disease Progression | Appointment 0, and 3, 6, 9 and 12 months after appointment 0

SECONDARY OUTCOMES:
Progression of the LCQ (Leicester Cough Questionnaire) | Appointment 0, and 3, 6, 9 and 12 months after appointment 0
Progression of the SOBQ (Shortness of Breath Questionnaire) | Appointment 0, and 3, 6, 9 and 12 months after appointment 0
Proportion of the Participants With Exacerbations | Appointment 0, and 3, 6, 9 and 12 months after appointment 0
Cases Of Death (All, Idiopathic Pulmonary Fibrosis Associated) | Up to 12 months
Proportion of the Participants, who After the 3 Week Titration Phase Receive the Full Maintenance Dosage Of Pirfenidone | 3, 6, 9 and 12 months after appointment 0
Dosage of Pirfenidone | Up to 12 months
Proportion of the Participants who Change the Dosage Of Pirfenidone | Up to 12 months
Reasons for the Dosage Change | Up to 12 months
Reasons for the Beginning, Change or Discontinuation of a Treatment of Comorbidities of Pirfenidone Associated Adverse Drug Reactions | Up to 12 months
Number of Participants With at Least one Adverse Drug Reaction Under the Therapy With Pirfenidone | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Germany (17):
  - Praxis Dr. med. Mathias Rolke und Dr. med. Peter Rückert, Aschaffenburg
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Dr. med. Martin Hoster, Dr. Hans-G. Lange von Stocmeier, Michael Behn und w., Bochum
  - Praxis Dr. med. Wilhelm Ammenwerth, Bochum
  - Augusta Kranken-Anstalt gGmbH, Bochum
  - Kliniken der Stadt Köln gGmbH Krankenhaus Merheim, Cologne
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Klinikum Werra-Meißner GmbH, Eschwege
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Universitätsklinikum Freiburg, Abteilung Pneumologie, Freiburg im Breisgau
  - Klinikum Fulda gAG; Universitätsmedizin Marburg, Campus Fulda, Fulda
  - Ev. Krankenhaus Göttingen-Weende E.V., Göttingen
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Universitätsklinikum Magdeburg Klinik für Kardiologie Angiologie u.Pneumologie, Magdeburg
  - Thoraxzentrum, Abt. Pneumologie, Münnerstadt
  - Praxis Dr. med. Matthias Waltert, Münster
  - Facharztzentrum üBAG, Sonneberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schreiber J, Schutte W, Koerber W, Seese B, Koschel D, Neuland K, Grohe C. Clinical course of mild-to-moderate idiopathic pulmonary fibrosis during therapy with pirfenidone: Results of the non-interventional study AERplus. Pneumologie. 2024 Apr;78(4):236-243. doi: 10.1055/a-2267-2074. Epub 2024 Apr 12. PMID 38608658